CLINICAL TRIAL: NCT02338674
Title: Combination Therapy of Tenofovir and Telbivudine in Immune-tolerant Patients With Chronic Hepatitis B Awaiting Assisted Reproduction
Brief Title: TDF and LdT in Immune-tolerant CHB Patients Awaiting Assisted Reproduction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Dongliang Li, Director, Department of Hepatobiliary Disease, Fuzhou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBV-AR
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; Telbivudine; Combined Modality Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COM (Experimental): COM group receives combination therapy of tenofovir and telbivudine (TDF and LdT) for at least 48 weeks
  Interventions: Drug: Tenofovir and telbivudine
- TDF (Active Comparator): TDF group receives single therapy of tenofovir (TDF) for at least 48 weeks
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir and telbivudine — tenofovir and telbivudine administered at least 48 weeks
  Other Names: combination therapy
  Arms: COM
Drug: Tenofovir — tenofovir administered at least 48 weeks
  Other Names: single therapy
  Arms: TDF

SUMMARY:
Immune-tolerant patients with chronic hepatitis B (CHB) awaiting assisted reproduction (AR) are required to initiate antiviral therapy due to laboratory safety. Additionally, rapid virus elimination is suggested to faciliate timely performance of AR. However, no consensus is reached regarding the antiviral therapy in this group. This study aimed to explore the efficacy and safety of tenofovir (TDF) and telbivudine (LdT) in this population.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years old with artificial reproductive needs
* Liver function (ALT) <40U/L for male and <30 for female
* HBV-DNA> 10e+5
* HBVeAg +
* History> 0.5 years

Exclusion Criteria:

* Cirrhosis
* Combined with other liver diseases such as autoimmune liver disease, alcoholic liver disease, fatty liver
* Liver or other parts of malignancies
* Bilirubin> 17.1
* GGT> 2ULN
* Liver transplant patients
* combined HCV, HDV, HIV infection
* A history of anti-HBV drug resistance
* History of habitual abortion
* previous fetal malformation history
* CRP> 3.0ng / ml
* Uncontrolled hypertension
* Proteinuria or Calculated creatinine clearance < 70 mL/min
* Heart failure or acute coronary syndrome
* Coagulopathy
* Drug or alcohol addiction
* Hyperlipidemia LDL> 4.6 or TG> 2.0
* Alphafetoprotein > 50 ng/mL
* Received interferon (pegylated or not) therapy within 6 months of the screening visit
* Evidence of hepatocellular carcinoma
* Received solid organ or bone marrow transplantation
* Was currently receiving therapy with immunomodulators (eg, corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents
* Known hypersensitivity to the study drugs, the metabolites, or formulation excipients

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With HBV DNA < 500 Copies/mL at Week 12 | week 12

SECONDARY OUTCOMES:
Percentage of Participants With HBV DNA < 500 Copies/mL at Week 24, 36 and 48 | Week 24, 36 and 48
Number of Participants With Normal Alanine Aminotransferase (ALT) at Week 12, 24, 36 and 48 | Week 12, 24, 36 and 48
Number of Participants With Hepatitis B e Antigen (HBeAg) Loss at Week 12, 24, 36 and 48 | Week 12, 24, 36 and 48
Number of Participants With Seroconversion to Antibody Against HBeAg (AntiHBe) at Week 12, 24, 36 and 48 | Week 12, 24, 36 and 48
Number of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 12, 24, 36 and 48 | Week 12, 24, 36 and 48
Number of Participants With Seroconversion to Antibody to HBsAg (AntiHBs) at Week 12, 24, 36 and 48 | Week 12, 24, 36 and 48
Occurrence of HBV Resistance Mutations | Baseline to Week 48
off-treatment recurrence of HBV | Week 72 to 96
Down syndrome Occurrence | week 13 of pregnancy
Fetal Malformations Occurrence | week 26 of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Dongliangli Li, Dr., Study Chair — Department of Hepatobiliary Disease
Locations (1):
- Fuzhou General Hospital, Xiamen Univ, Fuzhou, Fujian, China